CLINICAL TRIAL: NCT07120464
Title: Clinical Study on Immunogenicity and Safety of Lyophilized Vero Cell-Derived Human Rabies Vaccine in Special Populations
Status: Recruiting | Type: Observational
Sponsor: Liaoning Chengda Biotechnology CO., LTD (Industry)
Collaborators: Shenzhen Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Other Study IDs: CDB-RV-PM-2025001
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Rabies Exposure; Immunocompromised; Chronic Disease
Keywords: Immunocompromised Patients; Chronic Diseases; Elderly Population; Rabies Vaccine; Vaccine Immunogenicity
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy Adult Control Group: Healthy adults aged 18 to under 60 years who seek medical attention after confirmed WHO category II or III rabies exposure and have no known chronic illness or immunocompromising condition.
  Interventions: Other: Observation Only
- Immunocompromised Group: Participants diagnosed with rabies category II or III exposure who are immunocompromised due to conditions such as primary immunodeficiency, hematologic or solid malignancies, aplastic anemia, or autoimmune diseases receiving long-term immunosuppressive therapy. A total of 50 participants will be enrolled in this group.
  Interventions: Other: Observation Only
- Chronic Disease Group: Participants diagnosed with rabies category II or III exposure who have chronic health conditions including diabetes, chronic hepatitis, cirrhosis, chronic glomerulonephritis, nephrotic syndrome, or chronic renal insufficiency. A total of 50 participants will be enrolled in this group.
  Interventions: Other: Observation Only
- Elderly Group: Participants aged 60 years and above (including those aged exactly 60) with category II or III rabies exposure and no exclusionary comorbidities beyond age-related health changes. A total of 50 participants will be enrolled in this group.
  Interventions: Other: Observation Only

INTERVENTIONS:
Other: Observation Only — All participants will receive post-exposure rabies vaccination using either the Zagreb or Essen regimen, in accordance with national immunization guidelines.

SUMMARY:
This study adopts a parallel-controlled design and includes a study group and a control group. The study group will enroll 150 special population participants (including non-HIV-related immunocompromised individuals, patients with chronic diseases, and elderly individuals) who receive their first post-exposure treatment following WHO category II or III rabies exposure. The control group will include 30 healthy adults with similar exposure.

Blood samples will be collected at Day 14 and Day 90 after completion of the full vaccination schedule to assess rabies virus neutralizing antibody seroconversion rates and titers. Immunogenicity and antibody persistence will be compared between the two groups. Additionally, all adverse events occurring within 30 minutes and within 7 days after each dose will be recorded to evaluate safety.

DETAILED DESCRIPTION:
This is a controlled study consisting of a study group and a control group. The study group will include special population participants (non-HIV-related immunocompromised individuals, patients with chronic diseases, and elderly individuals) who are receiving their first clinical visit after confirmed WHO category II or III rabies exposure. The control group will include healthy adults aged 18 to under 60 years who also present after similar exposure. The study group will be further divided into three subgroups based on the health status of the participants, with 50 individuals in each subgroup:

1. Immunocompromised group: including individuals with primary immunodeficiency diseases, hematologic or solid organ malignancies, aplastic anemia, and autoimmune diseases under long-term immunosuppressive therapy;
2. Chronic disease group: including patients with diabetes, chronic hepatitis, cirrhosis, chronic glomerulonephritis, nephrotic syndrome, and chronic renal insufficiency;
3. Elderly group: participants aged 60 years and above (including those aged exactly 60).

If a participant meets criteria for more than one subgroup (e.g., aged ≥60 years and also has immunodeficiency or a chronic disease), subgroup assignment will be prioritized based on disease condition: immunocompromised first, then chronic disease, and finally elderly, to ensure each participant is assigned to the most representative subgroup.

All participants (both in the study and control groups) may choose either the Zagreb regimen (2-1-1) or the Essen regimen (five-dose schedule) for post-exposure rabies vaccination. Adverse events occurring within 0-7 days after each vaccine dose will be collected via telephone follow-up to understand post-vaccination responses.

Blood samples will be collected at Day 14 after completion of the full vaccination schedule (i.e., Day 35 from first dose for Zagreb regimen and Day 42 for Essen regimen), and again at Day 90 (Day 111 and Day 118 from first dose for Zagreb and Essen, respectively). Rabies virus neutralizing antibodies will be tested and compared between groups to evaluate the immunogenicity of rabies vaccination in special populations after exposure. Safety data will also be analyzed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with WHO category II or III rabies exposure presenting at the study site for post-exposure prophylaxis and vaccination.
* Subjects planned to be included in the control group, aged 18 to less than 60 years old, healthy as confirmed by medical history, physical examination, and clinical judgment before vaccination.
* Subjects planned to be included in the study group who meet any of the following conditions:

  1. Long-term immunocompromised status due to conditions including, but not limited to: clinically confirmed primary immunodeficiency diseases; hematologic or solid organ malignancies; aplastic anemia; clinically confirmed autoimmune diseases with immunosuppressive therapy lasting 4 weeks or longer within the past 12 months prior to enrollment; history of splenectomy or other major immunologic organ removal; hematopoietic stem cell or solid organ transplantation within 2 years prior to enrollment.
  2. Clinically confirmed diabetes mellitus, chronic hepatitis, liver cirrhosis, chronic glomerulonephritis, nephrotic syndrome, or chronic renal insufficiency.
  3. Age 60 years or older.
* Subjects or their legally authorized representatives are able to understand the study requirements and procedures, voluntarily agree to participate, and sign the informed consent form.
* Subjects are able to comply with all planned follow-up visits and provide valid identification documents of themselves and/or their legally authorized representatives.

Exclusion Criteria:

* History of previous rabies vaccination.
* History of human immunodeficiency virus (HIV) infection.
* Other conditions deemed unsuitable for participation in the clinical study by the investigator.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study uses a parallel controlled design with two groups: a study group and a control group. The study group will enroll approximately 150 special population subjects who present for post-exposure prophylaxis after category II or III rabies exposure. These special populations include individuals with immunocompromised conditions excluding HIV infection, patients with chronic diseases, and elderly subjects. The control group will include approximately 30 healthy adults aged 18 to less than 60 years presenting for post-exposure prophylaxis after category II or III rabies exposure.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rabies virus neutralizing antibody (RVNA) seropositivity rate and antibody level at Day 14 after full vaccination | 14 days post completion of full vaccination.
  The proportion of subjects with rabies virus neutralizing antibody (RVNA) ≥ 0.5 IU/ml and the antibody titer level in serum at 14 days after completion of the full vaccination schedule.
Rabies virus neutralizing antibody (RVNA) seropositivity rate and antibody level at Day 90 after full vaccination | 90 days post completion of full vaccination.
  he proportion of subjects with RVNA ≥ 0.5 IU/ml and the antibody titer level in serum at 90 days after completion of the full vaccination schedule.

SECONDARY OUTCOMES:
Safety profile of rabies vaccine | Within 30 minutes and 7 days after each vaccine dose.
  Incidence of local (injection site) and systemic (non-injection site) adverse events/reactions within 30 minutes and up to 7 days after each vaccine dose, including serious adverse events and other adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Huang, Principal Investigator — Shenzhen Center for Disease Control and Prevention
Locations (1):
- Luohu District People's Hospital., Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No